CLINICAL TRIAL: NCT06327451
Title: Evaluate the Efficacy and Safety of Atorvastatin Combined With Temozolomide in the Treatment of Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Chunsheng Kang, Principal Investigator, Clinical Professor, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2024-YX-037-01
Record Dates: First submitted 2024-02-20; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Glioblastoma, IDH-wildtype
MeSH Terms: conditions — Glioblastoma | interventions — Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atorvastatin administrating group (Experimental): According to the clinical standard dose of lipid-lowering drugs, the subjects were enrolled in this study. After 2 weeks of glioma surgery, one tablet of liptor was taken orally every night on the basis of STUPP protocol.
  Interventions: Drug: Atorvastatin 20mg

INTERVENTIONS:
Drug: Atorvastatin 20mg — Liptor is a capsule in the form of 20 mg, once daily.

SUMMARY:
Glioblastoma (GBM) is the primary intracranial malignant tumor with the highest morbidity and mortality, and the 5-year survival rate is less than 10%. The number of primary diagnostic patients and deaths of GBM in China ranks first in the world every year, which seriously threatens people's life and health. At present, the clinical treatment strategy of maximum surgical resection combined with concurrent chemo- and radio-therapy and TTF treatment is still not satisfactory, and the median survival time of GBM patients is only 14.4 months. Statins inhibit cholesterol production with few side effects and are widely used for cholesterol control in patients with hyperlipidemia. In recent years, statins have shown good anti-tumor effect. Our previous study found that statins can block the malignant progression of glioma mediated by EGFR pathway. Therefore, the investigators report a clinical study protocol designed to evaluate the clinical efficacy of a comprehensive treatment strategy of atorvastatin (ATO) combined with temozolomide (TMZ) in primary and recurrent glioblastomas with high EGFR expression.

The investigators designed a multicenter, single-arm, double-blind, phase II clinical trial to evaluate the efficacy and safety of oral ATO combined with TMZ in EGFR-high expressing GBM. After informed consent was signed by the patient or authorized family members, the patients were treated with the current STUPP regimen and ATO (20mg, qn) orally. The patients were regularly followed up for 52 weeks after treatment. The primary endpoint was progression-free survival (PFS), which was defined as the time from the start of GBM surgery to tumor progression (recurrence) or death. The secondary end point was the rate of tumor control, which was defined as the proportion of patients with a complete response, a partial response, or a stable disease that had shrunk or remained stable for a given period of time. Safety will be assessed during the study by monitoring of regular MRI scans, laboratory tests (liver function, lipid profile, blood routine), electrocardiography, vital signs (blood pressure, pulse, temperature), and weight.

The results of this clinical trial will provide key information on whether the oral combination of atorvastatin and temozolomide prolongs PFS in EGFR-high GBM patients with efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old and < 60 years old, both sexes;
2. sufficient evidence of glioma by MRI scan;
3. According to the 2021 WHO latest classification, the molecular pathology of postoperative glioma samples was diagnosed as WHO 4 glioblastoma;
4. The immunohistochemical results of postoperative glioma samples showed that EGFR score was 3 (standard: 0 was negative, 1-3 was positive);
5. normal blood routine and liver function;
6. fully understand the nature of the trial and sign the informed consent;
7. be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures;
8. no serious diseases or accidents requiring surgery;
9. normal immune function.

Exclusion Criteria:

1. allergy to atorvastatin or its components;
2. concomitant use of clarithromycin, itraconazole, ritonavir, saquinavir, lopinavir, cyclosporine, rifampicin, efavirenz, digoxin, warfarin, oral contraceptives;
3. other tumors (except glioma), hematological diseases or other known multiple organ failure, history of myasthenia gravis, heart failure, cerebral hernia and other serious complications;
4. History of cardiac insufficiency, arrhythmia, retinopathy, acute hepatic porphyrin, hepatic and renal insufficiency, obesity, uncontrolled diabetes and other metabolic diseases;
5. abnormal liver function or liver disease, including uncontrolled hepatitis;
6. other diseases that might interfere with the study, as determined by 2 attending neurosurgeons;
7. patients enrolled in a clinical trial within the past 4 weeks;
8. pregnant or lactating patients;
9. patients with poor compliance who could not complete the treatment;
10. other conditions that made the patient ineligible for enrollment as determined by the study investigator;
11. patients with a history of HIV and/or HBV/HCV or presence of HIV/HCV;
12. patients with a history of tuberculosis or known existence of tuberculosis;
13. patients with severe infection or signs/symptoms of infection within 2 weeks before the first dose of study drug;
14. patients who received live attenuated vaccine within 4 weeks before the first dose of study drug;
15. patients with previous solid organ transplantation or hematopoietic stem cell transplantation.

Those who meet any of the above criteria will not be selected.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | the time from the start of GBM surgery to tumor progression (recurrence) or death, whichever came first, assessed up to 52 weeks
  progression-free survival
Overall survival | the time from the start of GBM surgery to the day of death from any cause, whichever came first, assessed up to 52 weeks
  Overall survival
Tumor control rate | Changes in tumor size before and after treatment, assessed up to 52 weeks
  Tumor control rate

SECONDARY OUTCOMES:
Hepatic burden of GBM patients after receiving atorvastatin administration | 1, 3, and 6 months after enrollment
  This outcome is evaluation of hepatic burden of GBM patients after receiving atorvastatin administration. Since participant is enrolled in this research, peripheral blood will be collected for testing ALT, AST, GGT, ALP, TP, ALB, GLB, A/G, TBIL, DBIL, and IBIL. The physiological parameters of these index are as follows: ALT: 0~40 U/L; AST: 0~40 U/L; GGT: 0~40 U/L; ALP: 40~110 U/L; TP: 65~85 g/L; ALB: 40~55 g/L; GLB: 20~40 g/L; A/G: 1.5~2.5: 1; TBIL: 0~23 μmol/L; DBIL: 0~8 μmol/L; IBIL: 1~14 μmol/L.
Percentage of participants with treatment-related adverse events | 1, 3, and 6 months after enrollment
  This outcome is evaluation of safety and tolerability during combination therapy of atorvastatin and STUPP protocol. Percentage of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Chunsheng Kang, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No
According to the clinical standard dose of lipid-lowering drugs, the subjects were enrolled in this study. After 2 weeks of glioma surgery, one tablet of liptor was taken orally every night on the basis of other treatments.